CLINICAL TRIAL: NCT01787487
Title: Evaluation of Ruxolitinib and Azacytidine Combination as a Therapy for Patients With Myelofibrosis and Myelodysplastic Syndrome/ Myeloproliferative Neoplasm
Brief Title: Ruxolitinib Phosphate and Azacytidine in Treating Patients With Myelofibrosis or Myelodysplastic Syndrome/Myeloproliferative Neoplasm
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-0737; NCI-2013-00704 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2012-0737 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2013-02-06; First posted 2013-02-08 (Estimated); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Myelodysplastic/Myeloproliferative Neoplasm, Unclassifiable; Myelofibrosis Transformation in Essential Thrombocythemia; Polycythemia Vera, Post-Polycythemic Myelofibrosis Phase; Primary Myelofibrosis
MeSH Terms: conditions — Myeloproliferative Disorders; Polycythemia Vera; Primary Myelofibrosis | interventions — Azacitidine; ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (MF patients) (Experimental): Patients with MF receive ruxolitinib phosphate PO BID on days 1-28. Beginning course 4, patients also receive azacytidine SC or IV for 5 days. Treatment repeats every 28 days for 15 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Azacitidine; Other: Laboratory Biomarker Analysis; Drug: Ruxolitinib Phosphate
- Arm II (MDS/MPN patients) (Experimental): Patients with MDS/MPN receive ruxolitinib phosphate and azacytidine as in Arm I.
  Interventions: Drug: Azacitidine; Other: Laboratory Biomarker Analysis; Drug: Ruxolitinib Phosphate

INTERVENTIONS:
Drug: Azacitidine — Given SC or IV
  Other Names: 5 AZC; 5-AC; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; U-18496; Vidaza
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Ruxolitinib Phosphate — Given PO
  Other Names: INCB-18424 Phosphate; Jakafi

SUMMARY:
This phase II trial studies how well ruxolitinib phosphate and azacytidine work in treating patients with myelofibrosis or myelodysplastic syndrome/myeloproliferative neoplasm. Ruxolitinib phosphate may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as azacytidine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving ruxolitinib phosphate and azacytidine may be an effective treatment for myelofibrosis or myelodysplastic syndrome/myeloproliferative neoplasm.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the efficacy of the combination of RUX (ruxolitinib phosphate) with AZA (azacytidine) in patients with myelofibrosis (MF) (primary myelofibrosis, post polycythemia vera myelofibrosis, or post essential thrombocythemia myelofibrosis [PMF, post- PV MF, or post - ET MF]) in achieving objective improvements in disease status.

II. To determine the efficacy of the combination of RUX + AZA in patients with myelodysplastic syndromes/myeloproliferative neoplasms (MDS/MPN) including chronic myelomonocytic leukemia (CMML), atypical chronic myeloid leukemia (breakpoint cluster region [BCR]-c-abl oncogene 1, non-receptor tyrosine kinase [ABL1] negative: aCML), and myelodysplastic syndromes/myeloproliferative neoplasms, unclassifiable (MDS/MPN-U), in achieving objective improvements in disease status.

SECONDARY OBJECTIVES:

I. To determine the safety of the RUX + AZA combination in patients with MF and MDS/MPN.

TERTIARY OBJECTIVES:

I. To explore time to response (TTR) and duration of response (DOR). II. To explore the effect of the combination on anemia and transfusion dependence in patients with MF and MDS/MPN.

III. To explore the impact of baseline mutational profile on International Working Group (IWG)-Myeloproliferative Neoplasms Research and Treatment (MRT) response and overall survival in patients with MF and MDS/MPN.

IV. To explore the impact of baseline anemia on overall survival in patients with MF and MDS/MPN.

OUTLINE: Patients are assigned to 1 of 2 treatment arms.

ARM I (MF): Patients with MF receive ruxolitinib phosphate orally (PO) twice daily (BID) on days 1-28. Beginning course 4, patients also receive azacytidine subcutaneously (SC) or intravenously (IV) for 5 days. Treatment repeats every 28 days for 15 courses in the absence of disease progression or unacceptable toxicity.

ARM II (MDS/MPN): Patients with MDS/MPN receive ruxolitinib phosphate and azacytidine as in Arm I.

After completion of study treatment, patients are followed up for 30 days and up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of primary myelofibrosis (PM), post polycythemia vera myelofibrosis (PPV MF), or post essential thrombocythemia myelofibrosis (PET MF) requiring therapy, including those previously treated and relapsed or refractory, or if newly diagnosed, with intermediate or high risk according to International Working Group (IWG-MRT) criteria
* Patients with a diagnosis of myelodysplastic syndrome/myeloproliferative neoplasm, unclassifiable (MDS/MPN-U) that require therapy
* Understanding and voluntarily signing an Institutional Review Board (IRB)-approved informed consent form
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2
* Direct bilirubin of =< 2 mg/dL
* Serum glutamate pyruvate transaminase (SGPT) =< 2.5 x upper limit of normal (ULN) or 5 x ULN if related to MF or MDS/MPN associated liver infiltration
* If total bilirubin is =< 2, fractionation is not required for eligibility determination
* Creatinine =< 2.5 mg/dL
* Platelets >= 50 x 10^9/L
* Absolute neutrophil count (ANC) >= 1.0 x 10^9/L

Exclusion Criteria:

* For the MF and MDS/MPN-U arms (arms 1 & 2), use of any other standard drug (except hydroxyurea, anagrelide, growth factors, Revlimid, clofarabine, etc) or experimental drug or therapy within 14 days of starting study therapy
* Patients previously treated with RUX or AZA (only applicable for the MF and MDS/MPN arms)
* Any serious psychological condition or psychiatric illness that would prevent the subject from signing the informed consent document, in the investigator opinion
* Pregnant or lactating females
* Subjects of childbearing potential who are unwilling to take appropriate precautions (from screening through follow-up) to avoid becoming pregnant or fathering a child; females of non-childbearing potential are defined as women who a) are 55 years of age with history of amenorrhea for 1 year OR b) are surgically sterile for at least 3 months; for females of childbearing potential, or for males, pregnancy must be avoided by taking appropriate precautions; these precautions and the methods of contraception should be communicated to the subjects and their understanding confirmed
* Any condition which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study
* Known positive for human immunodeficiency virus (HIV) or with known active infectious hepatitis, type A, B or C
* Patients with active malignancy of other type than required for this study, are not eligible with the exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast; patients with malignancies with indolent behavior such as prostate cancer treated with radiation or surgery can be enrolled in the study as long as they have a reasonable expectation to have been cured with the treatment modality received

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2013-03-13 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (complete remission, partial remission, clinical improvement) in patients with myelofibrosis | Up to 24 weeks
  The method of Thall, Simon and Estey will be used for futility monitoring for this study. The objective response rate will be estimated along with the Bayesian 95% credible interval.
Objective response rate (complete remission, partial remission, and hematologic improvement) in patients with myelodysplastic syndromes/myeloproliferative neoplasms | Up to 24 weeks
  The method of Thall, Simon and Estey will be used for futility monitoring for this study.

SECONDARY OUTCOMES:
Incidence of adverse events defined as grade 3-4 clinically relevant non-hematologic toxicity or a serious adverse event that is felt to be drug related as assessed by the Common Terminology Criteria for Adverse Events version 4.0 | Up to 30 days after completion of study treatment
  The method of Thall, Simon and Estey will be used for toxicity monitoring for this study.

CONTACTS AND LOCATIONS:
Overall Officials: Naval Daver, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Masarova L, Verstovsek S, Hidalgo-Lopez JE, Pemmaraju N, Bose P, Estrov Z, Jabbour EJ, Ravandi-Kashani F, Takahashi K, Cortes JE, Ning J, Ohanian M, Alvarado Y, Zhou L, Pierce S, Gergis R, Patel KP, Luthra R, Kadia TM, DiNardo CD, Borthakur G, Bhalla K, Garcia-Manero G, Bueso-Ramos CE, Kantarjian HM, Daver N. A phase 2 study of ruxolitinib in combination with azacitidine in patients with myelofibrosis. Blood. 2018 Oct 18;132(16):1664-1674. doi: 10.1182/blood-2018-04-846626. Epub 2018 Sep 5. PMID 30185431
- [Derived] Assi R, Kantarjian HM, Garcia-Manero G, Cortes JE, Pemmaraju N, Wang X, Nogueras-Gonzalez G, Jabbour E, Bose P, Kadia T, Dinardo CD, Patel K, Bueso-Ramos C, Zhou L, Pierce S, Gergis R, Tuttle C, Borthakur G, Estrov Z, Luthra R, Hidalgo-Lopez J, Verstovsek S, Daver N. A phase II trial of ruxolitinib in combination with azacytidine in myelodysplastic syndrome/myeloproliferative neoplasms. Am J Hematol. 2018 Feb;93(2):277-285. doi: 10.1002/ajh.24972. Epub 2017 Nov 27. PMID 29134664
- See also: MD Anderson Cancer Center — http://www.mdanderson.org